CLINICAL TRIAL: NCT06425497
Title: DE NOVO DONOR SPECIFIC ANTIBODIES AFTER KIDNEY TRANSPLANTATION: SINGLE-CENTER RETROSPECTIVE STUDY
Acronym: PTV-DSAaKT
Status: Completed | Type: Observational
Sponsor: University of Rome Tor Vergata (Other)
Responsible Party: Principal Investigator, Roberta Angelico, Associate Professor, University of Rome Tor Vergata
Other Study IDs: sperimentazioni PTV 92.24
Record Dates: First submitted 2024-05-17; First posted 2024-05-22 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Kidney Transplant; Complications; Immunosuppression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Kidney transplant patients: The study population will be composed by patients who underwent a kidney transplant, single or double, from a deceased or living donor, from 01/01/2010 to 07/31/2023 at the U.O.C. of the Hepatobiliary Surgery and Transplants of the Tor Vergata Polyclinic, with at least one year of post-transplant follow-up.
  Interventions: Other: The dosage of dnDSA

INTERVENTIONS:
Other: The dosage of dnDSA — Flow cytometric analysis using FlowPRA Screening Test and/or Luminex Single Antigen Beads class I and II- IgG (cut- positivity off = MFI> 1000)

SUMMARY:
To investigate the variations of Donor Specific Antibodies in kidney transplant patients based on the type of immunosuppressive therapy adopted and immunosuppressive blood levels.

DETAILED DESCRIPTION:
Retrospective observational monocentric study at the U.O.C. of Hepatobiliary Surgery and Transplants of Tor Vergata Polyclinic. All kidney transplant patients in the indicated study period will be enrolled and followed at the U.O.C. clinic.

For each patient, demographic, transplant and post-transplant data will be collected. In the latter, data relating to dnDSA will be registered, searching for a possible triggering cause at the anamnestic level.

The dosage of dnDSA is performed in common clinical practice in a routine manner in all patients undergoing kidney transplant, using the method "Flow cytometric analysis using FlowPRA Screening Test and/or Luminex Single Antigen Beads class I and II- IgG (cut- positivity off = MFI> 1000)".

The blood dosage of the immunosuppressor is measured during routine checks and a comparison is made between Tacrolimus-based immunosuppressive therapy and other immunosuppressive therapy, highlighting the differences in the risk of developing dnDSA and in graft and patient survival.

ELIGIBILITY:
Inclusion Criteria:

* Patients,both male and female over the age of 18
* Patients with at least one year of follow-up

Exclusion Criteria:

* Combined liver-kidney or pancreas-kidney transplants
* Re-transplants
* Patients with follow-up less than one year

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be composed by patients who underwent a kidney transplant, single or double, from a deceased or living donor, from 01/01/2010 to 07/31/2023 at the U.O.C. of the Hepatobiliary Surgery and Transplants of the Tor Vergata Polyclinic, with at least one year of post-transplant follow-up.
Sampling Method: Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2024-05-06 (Actual)

PRIMARY OUTCOMES:
Development of dnDSA in kidney transplant patients | • Pre-transplant • Baseline (I PODs) • At one week • At one month • At 3 months • At 6 months • At one year • At 5 years old • At 10 years old
  Define the incidence of development of dnDSA in patients undergoing kidney transplantation.

SECONDARY OUTCOMES:
Graft survival | 5 and 10 years
  Graft survival At 5 and 10 years
Patient survival | 5 and 10 years
  Patient survival at 5 and 10 years
Blood dosage levels of post-transplant immunosuppressive drugs | • At one week • At one month • At 3 months • At 6 months • At one year • At 5 years old • At 10 years old
  Blood dosage levels of post-transplant immunosuppressive drugs (tacrolemia, ciclosporinemia, everolemia, sirolemia);
Donor-recipient HLA mismatch | Pre-transplant
  Donor-recipient HLA mismatch

CONTACTS AND LOCATIONS:
Overall Officials: Roberta Angelico, MD, Principal Investigator — University of Rome Tor Vergata